CLINICAL TRIAL: NCT04368403
Title: A Phase 1, Open-label, Multiple-dose Study of KHK4827 in Subjects With Systemic Sclerosis
Brief Title: A Study of KHK4827 in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4827-007
Record Dates: First submitted 2020-04-13; First posted 2020-04-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; brodalumab; KHK4827
MeSH Terms: conditions — Scleroderma, Systemic | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KHK4827 (Experimental)
  Interventions: Drug: KHK4827

INTERVENTIONS:
Drug: KHK4827 — 210 mg every 2 weeks (Q2W), subcutaneous (SC) injection

SUMMARY:
Exploratory evaluation of pharmacokinetics and safety of KHK4827 in subjects with systemic sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the criteria for diagnosis of the Diagnostic Criteria, Severity Classification, and Clinical Practice Guidelines for Systemic Sclerosis （Japanese Dermatological Association 2016） at the pre-examination
* Subject presented the first symptoms of sclerosis other than Raynaud's phenomenon within 60 months before enrollment
* Subject who has systemic sclerosis accompanied by moderate to severe skin thickening with an mRSS of 10 to <30 at the pre-examination and who has progressing skin thickening

Exclusion Criteria:

1. Any of the following significant concomitant diseases:

   * Type 1 diabetes
   * Poorly controlled type 2 diabetes (HbA1c > 8.5%)
   * Congestive heart failure (Class II to IV of the New York Heart Association Functional Classification)
   * Myocardial infarction, unstable angina, or stroke occurring within 12 months before the first dose of investigational product
   * Poorly controlled hypertension (systolic pressure > 150 mm Hg or diastolic pressure > 90 mg Hg at screening)
   * Severe chronic lung disease (%Forced Vital Capacity (FVC) < 60% and %Diffusing capacity of lung for carbon monoxide (DLco) < 40%, calculated according to the Reference Values for Spirometry, Including Viral Capacity, in Japanese Adults Calculated with the LMS Method and Compared with Previous Values [Japanese Respiratory Society])
   * Major chronic inflammatory diseases or connective tissue diseases other than scleroderma
2. Patient has a history or evidence of a psychiatric disorder, alcohol and/or substance abuse, or any other mental health disorder that, in the opinion of the investigators, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
3. Patient has a history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at enrollment
4. Patient has severe depression based on a total score of ≥ 15 on the Patient Health Questionnaire-8 (PHQ-8) at enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
serum KHK4827 concentration | Pre-dose, Week 1, 2, 4, 8, 12, 16, 22, 24, 36, 48, 52 and every 24 weeks through study completion until 2025.

SECONDARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) from baseline | Pre-dose, Week 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and every 8 weeks through study completion until 2025.
  mRSS: scored 0(normal), 1(mild), 2(moderate), or 3(severe) per each site, assessed in 17 different body sites, total score=51

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tokyo Hospital, Bunkyo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.
URL: https://vivli.org/ourmember/kyowa-kirin/

REFERENCES:
- [Derived] Fukasawa T, Yoshizaki A, Ebata S, Fukayama M, Kuzumi A, Norimatsu Y, Matsuda KM, Kotani H, Sumida H, Yoshizaki-Ogawa A, Kagebayashi H, Sato S. Interleukin-17 pathway inhibition with brodalumab in early systemic sclerosis: Analysis of a single-arm, open-label, phase 1 trial. J Am Acad Dermatol. 2023 Aug;89(2):366-369. doi: 10.1016/j.jaad.2023.02.061. Epub 2023 Mar 29. No abstract available. PMID 36997069